CLINICAL TRIAL: NCT01502644
Title: Opioid Treatment for Chronic Low Back Pain and the Impact of Mood Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Arthritis Foundation (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ajay D. Wasan,M.D.,M.Sc., Assistant Professor of Anesthesiology and Psychiatry, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007P-001047; 5K23DA020681-05 (NIH)
Record Dates: First submitted 2011-12-28; First posted 2012-01-02 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Chronic Low Back Pain; Degenerative Disc Disease; Depression; Anxiety
Keywords: low back pain; opioids; mood symptoms
MeSH Terms: conditions — Intervertebral Disc Degeneration; Depression; Anxiety Disorders; Low Back Pain | interventions — Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: During the first 2 weeks of treatment participants took short-acting morphine or oxycodone for 1 week and placebo for 1 week in random order. Participants and investigators were blinded during this period. The remainder of the study was conducted in an open-label design.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Negative Affect (NA) (Active Comparator): Participants with low NA (HADS score ≤5 on each subscale) received placebo or active opioid drug (immediate-release morphine 15 to 30 mg or oxycodone 5 to 10 mg) up to three times a day as needed for 1 week each in random order, followed by morphine or oxycodone titrated to a maximum allowable daily dose in morphine equivalents of 30 mg for short-acting medication and 60 mg for long-acting medication, respectively, three times a day for up to 20 weeks, followed by morphine or oxycodone tapering (individualized opioid dose was decreased by approximately 25% each week) for 4 weeks.
  Interventions: Drug: Oxycodone; Drug: Morphine; Drug: Placebo
- Moderate NA (Active Comparator): Participants with moderate NA (HADS score ≥6 to ≤8 on each subscale) received placebo or active opioid drug (immediate-release morphine 15 to 30 mg or oxycodone 5 to 10 mg) up to three times a day as needed for 1 week each in random order, followed by morphine or oxycodone titrated to a maximum allowable daily dose in morphine equivalents of 30 mg for short-acting medication and 60 mg for long-acting medication, respectively, three times a day for up to 20 weeks, followed by morphine or oxycodone tapering (individualized opioid dose was decreased by approximately 25% each week) for 4 weeks.
  Interventions: Drug: Oxycodone; Drug: Morphine; Drug: Placebo
- High NA (Active Comparator): Participants with high NA (HADS score ≥9 on each subscale) received placebo or active opioid drug (immediate-release morphine 15 to 30 mg or oxycodone 5 to 10 mg) up to three times a day as needed for 1 week each in random order, followed by morphine or oxycodone titrated to a maximum allowable daily dose in morphine equivalents of 30 mg for short-acting medication and 60 mg for long-acting medication, respectively, three times a day for up to 20 weeks, followed by morphine or oxycodone tapering (individualized opioid dose was decreased by approximately 25% each week) for 4 weeks.
  Interventions: Drug: Oxycodone; Drug: Morphine; Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone — Daily dosage up to 120 mg
Drug: Morphine — Daily dosage up to 90 mg immediate release or 180 mg extended release
  Other Names: Morphine sulfate (MS) Contin; Morphine sulfate instant release (MSIR); Morphine sulfate extended release (MSER)
Drug: Placebo — Placebo-matching oxycodone, placebo-matching morphine

SUMMARY:
Opioids are frequently prescribed for chronic low back pain (CLBP). Psychiatric illness, such as high levels of depression and anxiety symptoms, is a common co-occurrence in chronic pain patients (and is termed comorbid negative affect [NA]). The purpose of the study is to determine whether CLBP patients with either a high vs. a low or moderate degree of NA have different pain relief responses to oral opioids.

DETAILED DESCRIPTION:
The level of high, moderate or low NA was determined based on the participant's score on the Hospital Anxiety and Depression Scale (HADS). The HADS is a self-reported questionnaire that has 14 questions related to 2 domains: Anxiety subscale (7 questions) and Depression subscale (7 questions). Each item on the questionnaire is scored from 0 (least amount of anxiety/depression) to 3 (greatest amount of anxiety/depression), with total score between 0 and 21 for either anxiety or depression. Participants were assigned to high, moderate or low NA groups using the following HADS score criteria:

* High NA = HADS score ≥9 on each subscale
* Moderate NA = HADS score ≥6 to ≤8 on each subscale
* Low NA = HADS score ≤5 on each subscale

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain > 3/10
* Pain > 1 year
* Degenerative disc disease as seen on magnetic resonance imaging (MRI), which must meet minimum disc grading criteria: at least a grade III disc degeneration, a hyperintense zone, or abnormal disc morphology.
* Patients who may have had back surgery will be included.
* No epidural steroids or other nerve blocks for back pain either two weeks before or during the study period.
* No opioids or on short-acting opioids only (max. daily amount=120 mg morphine equivalents). It is not feasible to recruit only opioid naive patients.
* Must agree to 2-week washout for those on opioids.
* No active substance abuse.
* No intention to take new pain or psychiatric treatments during the study, including chiropractic, physical therapy, or complementary or alternative treatments (CAM). It is not feasible to take participants off of any other pain medications, such as nonsteroidal anti-inflammatory drugs (NSAIDS).
* No pregnancy or the intent to become pregnant during the study, and no nursing mothers.
* Women, who are able to bear children, must agree to use contraceptives throughout the study.
* In men, normal baseline testosterone levels.

Exclusion Criteria:

* Patients with pain due to disorders not including a component of disc degeneration, or those with unknown causes of pain will be excluded.
* Patients with the intent to undergo back surgery will be excluded.
* Patients with a history of recent or ongoing alcohol or other drug addiction disorders will be excluded.
* Patients with any history of substance abuse of opioids will be excluded.
* Patients whose diagnosis cannot be firmly established according to criteria described above would not be included.
* Patients whose medical and psychiatric comorbidities are not well controlled, or who are currently experiencing an acute exacerbation of the medical comorbidity, will be excluded.
* Males with abnormal testosterone levels will be excluded (normal range is 1800-6650 pg/ml).
* Female patients who nursing will be excluded.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay D Wasan, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers with chronic low back pain (CLBP) and psychiatric illness (comorbid negative affect [NA]) were recruited to participate in this trial.
Pre-assignment Details: NA level determined by Hospital Anxiety and Depression Scale (HADS) score: Anxiety and Depression subscales with 7 questions each, each question scored 0 (least) to 3 (greatest) amount of anxiety/depression, total score 0-21. High NA=score ≥9 on each subscale, Moderate NA=score ≥6 to ≤8 on each subscale, Low NA=HADS score ≤5 on each subscale.
Groups:
- Enrolled at Visit 1: All participants who satisfied pre-screening requirements and were enrolled at Visit 1.
- Low NA: Participants with low NA (HADS score ≤5 on each subscale) received placebo or active opioid drug (immediate-release morphine 15 to 30 mg or oxycodone 5 to 10 mg) up to three times a day as needed for 1 week each in random order, followed by morphine or oxycodone titrated to a maximum allowable daily dose in morphine equivalents of 30 mg for short-acting medication and 60 mg for long-acting medication, respectively, three times a day for up to 20 weeks, followed by morphine or oxycodone tapering (individualized opioid dose was decreased by approximately 25% each week) for 4 weeks.
Period: Enrolled at Visit 1 After Pre-screening
Arm/Group | Enrolled at Visit 1 | Low NA | Moderate NA | High NA
Started | 81 | 0 | 0 | 0
Completed | 72 (Participants who completed Visit 1 were assigned to 1 of the 3 NA groups for remainder of the trial) | 0 | 0 | 0
Not Completed | 9 | 0 | 0 | 0
Not completed — Illegal Drugs in Urine Drug Test | 1 | 0 | 0 | 0
Not completed — History of Opioid Substance Use Disorder | 2 | 0 | 0 | 0
Not completed — Declined to Participate further | 6 | 0 | 0 | 0
Period: Assigned to NA Groups
Arm/Group | Enrolled at Visit 1 | Low NA | Moderate NA | High NA
Started | 0 | 30 | 10 | 32
Completed | 0 | 24 (Completed = completed at least 50% of the opioid treatment period (at least 10 weeks of treatment)) | 7 (Completed = completed at least 50% of the opioid treatment period (at least 10 weeks of treatment)) | 24 (Completed = completed at least 50% of the opioid treatment period (at least 10 weeks of treatment))
Not Completed | 0 | 6 | 3 | 8
Not completed — Drop Out due to Side Effects | 0 | 6 | 2 | 7
Not completed — Illegal Drugs in Urine Drug Test | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population, all participants who completed at least 50% of the opioid treatment period (at least 10 weeks of treatment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Low NA | Moderate NA | High NA | Total
Number analyzed (Participants) | 24 | 7 | 24 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.9) | 54 (11.7) | 49 (12.2) | 51.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 14 | 33
  Male | 8 | 4 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Average Daily Pain Score
Description: Participants rated their average lower back pain over the past 24 hours using an 11-point scale (0=no pain to 10=worst possible pain) and recorded it in an electronic diary. The percent change in pain score from baseline is calculated using weekly averages for up to 20 weeks. Linear mixed modeling (LMM) analysis was used to allow for inclusion in the analysis of the majority of participants with any missing data. For the LMM model, group, group × week, average baseline pain, and opioid use at baseline (yes/no) were entered as fixed effects using an autoregressive covariance structure. Participant, intercept, and week were entered as random effects, using a compound symmetry covariance structure. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 20
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Low NA | Moderate NA | High NA
Number analyzed (Participants) | 24 | 7 | 24
percent change | 38.6 (35.0) | 30.0 (24.4) | 20.6 (26.5)
Statistical Analysis 1: Comparison: Low NA vs High NA; Test type: Other; p = 0.01, Linear Mixed Modeling; Group, group×week, average baseline pain, and opioid use at baseline were entered as fixed effects using an autoregressive covariance structure; Mean Difference (Net) = 18.0, 95% CI 2-sided [3.7 to 32.2]

ADVERSE EVENTS:
Description: Adverse events were not collected for this study.
Arm/Group | Low NA | Moderate NA | High NA
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/10 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes